CLINICAL TRIAL: NCT05250310
Title: The Effect of Structured Lifestyle Modification and Yoga Practice on Metabolic Processes Associated With Cardiovascular Disease
Acronym: SLYM II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have closed the study as subjects were not interested in participating.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Annapoorna Kini, Director, Cardiac Catheterization Laboratory, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 15-2147
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; metabolic abnormality; chair yoga; micro RNA
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Two group randomization 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga (Active Comparator): Patients randomized to Yoga arm will practice chair yoga for 30 minutes at least three days a week for 16 weeks
  Interventions: Behavioral: Chair Yoga
- Standard of Care (No Intervention): Control group patients will follow standard of care (SOC) treatment.

INTERVENTIONS:
Behavioral: Chair Yoga — Yoga poses performed in a chair
  Arms: Yoga

SUMMARY:
The aim of the prospective randomized single center study is to evaluate the effect of a short-term (16 weeks) yoga program on micro RNA (miRNA) expression and cardiovascular disease (CVD) risk factors in patients with CVD.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) and metabolic syndrome (MetS) are major public health problems in the USA and worldwide. Yoga has been proven effective in numerous studies to improve cardiovascular risk factors, with a reduction in the risk of heart attacks and strokes. MicroRNAs (miRNAs) have recently emerged as key regulators of metabolism by playing a crucial role in cholesterol and lipid metabolism, fatty acid metabolism, insulin and glucose homeostasis. Yoga has been shown to induce a dynamic shift in miRNAs and reset their target genes expression associated with metabolites and pathways connected to CVD and MetS to a normal physiological state. 120 subjects will be included in the study. After recruitment, subjects will be randomized to one of two groups: Yoga (n=60) or Control (n=60) group. Patients randomized to Yoga, will practice yoga poses in a chair for 30 min at least 3 days a week by watching video instruction for 16 weeks. Control group patients will follow standard of care (SOC) treatment. At the enrollment day and at the 16-weeks follow-up visit, 15ml of blood will be collected from all participants for miRNAs expression profile.

ELIGIBILITY:
Inclusion criteria:

* Subjects eligible for the study are 18-80 year old adults.
* Underwent percutaneous coronary intervention (PCI) at the catheterization lab of Mount Sinai Hospital (New York, New York) or have non-obstructive coronary artery disease and at least one CVD risk factor (hypertension, hypercholesterolemia, diabetes mellitus, or obesity) or metabolic abnormality (fasting plasma glucose ≥ 100 mg/dl, documented previous diagnosis of hypertension, serum triglycerides ≥ 150 mg/dl, or HDL cholesterol < 40 mg/dl).
* Subjects diagnosed with metabolic syndrome, which is defined as three or more of the following conditions: (1) Central or abdominal obesity (waist circumference > 40 inches for men and > 35 inches for women); (2) High triglycerides (≥150 mg/dL or triglycerides treatment); (3) Low HDL cholesterol (<40 mg/dL for men and <50 mg/dL for women) or low HDL-C treatment; (4) High blood pressure (≥130/85 mmHg) or antihypertensive medications; (5) High fasting glucose (≥100 mg/dL) or type 2 diabetes mellitus.
* Participants must be able to willingly consent to study participation and must be able to comply with the study requirements.

Exclusion Criteria:

* Physical/psychological limitation or unwillingness to practice yoga,
* Congestive heart failure, known arrthymias or prior Automated Implantable Cardioverter-Defibrillator /pacemaker or any metallic implants,
* Rheumatological/immunological diseases,
* History of transplant,
* Moderate to severe chronic obstructive pulmonary disease, debilitating or severe systemic Illness,
* Subjects who are pregnant or postpartum less than 6 months,
* Liver disease or alcohol use of more than 7 alcoholic drinks/week in women and more than 14 drinks/week in men

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
micro RNA expression | End of study, at 22 months

SECONDARY OUTCOMES:
Body weight | End of study, at 22 months
  Body weight, kg
Waist circumference | End of study, at 22 months
  Waist circumference, inches
Blood pressure | End of study, at 22 months
  blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No